CLINICAL TRIAL: NCT02240134
Title: Wood Stove Interventions and Child Respiratory Infections in Rural Communities
Brief Title: Wood Stove Interventions and Child Respiratory Health
Acronym: KidsAIR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Montana (Other)
Collaborators: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Responsible Party: Principal Investigator, Curtis Noonan, Principal Investigator, Professor, University of Montana
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRB 276-13; R01ES022649 (NIH)
Record Dates: First submitted 2014-09-10; First posted 2014-09-15 (Estimated); Results first posted 2022-06-02 (Actual); Last update posted 2022-06-22 (Actual); Status verified 2022-06

CONDITIONS: Lower Tract Respiratory Infection

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Education Intervention (Tx1) (Experimental): The education components for this intervention are based on recent observations and recommendations from tribal, local, state and federal agencies. The intervention will be a combination of a strong education campaign coupled with the distribution of inexpensive tools to the homes that will enable the residents to burn wood more efficiently.
  Interventions: Behavioral: Education Intervention (Tx1)
- Air Filtration Unit Treatment (Tx2) (Active Comparator): Within each randomly assigned home, a 20" x 18" Filtrete air filtration unit (Ultra Clean Air Purifiers, 3M, St. Paul, MN) will be placed in the same room as the wood stove.
  Interventions: Device: Air Filtration Unit Treatment (Tx2)
- Placebo Intervention (Tx3) (Sham Comparator): Similar to Tx1, a 20" x 18" Filtrete air filtration unit will be installed within the wood stove home. Instead of a high efficiency filter, the units will utilize a placebo filter.
  Interventions: Device: Placebo Intervention (Tx3)

INTERVENTIONS:
Behavioral: Education Intervention (Tx1) — The intervention will be a combination of a strong education campaign coupled with the distribution of inexpensive tools to the homes that will enable the residents to burn wood more efficiently.
  Arms: Education Intervention (Tx1)
Device: Air Filtration Unit Treatment (Tx2) — A 20" x 18" Filtrete air filtration unit (Ultra Clean Air Purifiers, 3M, St. Paul, MN) will be placed in the same room as the wood stove. These units are rated by their ability to provide an equivalent amount of contaminant free air into the space, and have a smoke Clean Air Delivery Rate of 112. The electrostatically charged filters in these units are approximately 85% efficient at removing 0.2 micron particles (cigarette smoke size particles) and over 95% efficient at removing 3 micron particles. The unit will be operated on the "high" setting throughout the duration of the six-month assessment winter periods. Filters will be changed out by the Community Coordinator approximately once per month in an effort to maximize collection efficiency.
  Arms: Air Filtration Unit Treatment (Tx2)
Device: Placebo Intervention (Tx3) — Similar to Tx1, a 20" x 18" Filtrete air filtration unit will be installed within the wood stove home. Instead of a high efficiency filter, the units will utilize a placebo filter.
  Arms: Placebo Intervention (Tx3)

SUMMARY:
Acute lower respiratory tract infections (LRTIs) account for more than 27% of all hospitalizations among US children under five years of age, with recurrent LRTIs in children a recognized risk factor for asthma. Residential biomass combustion leads to elevated indoor levels of fine particulate matter (PM2.5) that often exceed current health-based air quality standards. PM2.5 exposure is associated with many adverse health outcomes, including a greater than three-fold increased risk of LRTIs. To date, exposure reduction strategies in wood stove homes have been either inconsistently effective or include factors that limit widespread dissemination and continued compliance in rural and economically disadvantaged populations. In this project, the investigators propose to test the efficacy of two intervention strategies for reducing indoor wood smoke PM2.5 exposures and children's risk of LRTI in three unique and underserved settings: (1) rural mountain valley communities in western Montana; (2) Navajo Nation communities; and (3) Alaska Native Villages. The investigators will conduct a three-arm randomized placebo-controlled post-only intervention trial in wood stove homes with children less than five years old. Education on best-burn practices and training on the use of simple instruments (i.e., stove thermometers and wood moisture meters) will be introduced as one intervention arm (Tx1). This intervention will be evaluated against an indoor air filtration unit arm (Tx2), as well as a placebo arm (Tx3, sham air filters). The primary outcome will be LRTI incidence among children under five years of age. To allow for detection of exposure and outcome differences within each of the three regions, a sample of 324 homes, or 108 within each study area will be equally assigned to each of the three intervention arms. The overall hypothesis is that a low-cost, educational intervention targeting indoor wood smoke PM2.5 exposures will be sustainable, and can reduce children's risk of LRTI in underserved Native and rural communities.

DETAILED DESCRIPTION:
Rural and Native areas of the western United States (US) and Alaska experience substantial exposure and health disparities compared to more populated urban centers. One such source of disparity is the elevated inhalation exposures related to the use of wood stoves for home heating. Within rural areas of Montana, Alaska, and the Navajo Nation, research has shown that residential biomass combustion leads to indoor levels of fine particulate matter (PM2.5) that often exceed current health-based air quality standards. Parallel findings have been observed in several developing countries where biomass combustion is commonly used for cooking and/or heating. This is concerning, as PM2.5 exposure is associated with many adverse health outcomes, including a greater than three-fold increased risk of acute respiratory tract infections. Throughout the world, lower respiratory tract infections (LRTIs) are the most common cause of death in children under five years of age, and account for more than 27% of all hospitalizations among US children under five years. Importantly, untoward effects of recurrent LRTIs are cumulative in children and a recognized risk factor for asthma.

Currently, there is a global effort to reduce indoor biomass smoke exposures in developing countries. A recent intervention trial found that exposure reductions following the introduction of improved cookstoves was protective for severe infant pneumonia. Similar evidence-based efforts are warranted in rural and Native American communities in the US that suffer from elevated rates of childhood LRTI and commonly use wood for residential heating. The investigators have previously demonstrated that a community-wide wood stove changeout program (i.e., replacing old wood stoves with newer model wood stoves) resulted in reduced wintertime ambient PM2.5 and corresponding reductions in occurrence of childhood wheeze and respiratory infections. In this and other studies, however, inconsistent effects on indoor air quality following the introduction of newer technology wood stoves have been observed. The investigators have also shown that the introduction of air filtration units is a less costly and more efficacious strategy for reducing indoor wood smoke exposures. Nevertheless, the energy costs of operation and need for filter replacement (maintenance) remain barriers to widespread dissemination and continued compliance in rural and economically disadvantaged communities. Experience with these interventions and qualitative input from wood stove experts suggest that educational interventions related to wood stove operation can translate to low-cost and sustainable strategies that reduce indoor biomass combustion exposures and improve respiratory health.

In this project, the investigators propose to test the efficacy of an education-based intervention strategy for reducing indoor wood smoke exposures and children's risk of LRTI in three unique and underserved settings. This study is a three-arm randomized trial in wood stove homes with children less than five years old. Education on best-burn practices and training on the use of simple instruments (i.e., stove thermometers and wood moisture meters) will be introduced as one intervention arm (Tx1). This intervention will be evaluated against an indoor air filtration unit arm (Tx2), as well as a placebo arm (Tx3, sham air filters). The primary outcome will be LRTI incidence among children under five years of age. A sample of 324 homes, or 108 within each study area equally assigned to each of the three intervention arms, will allow for detection of exposure and outcome differences within each of the three regions. Through three Aims, the overall hypothesis is that a low-cost, educational intervention targeting indoor wood smoke (PM2.5) exposures will be an effective, sustainable strategy for reducing children's risk of LRTI in underserved Native and rural communities.

Aim 1: Compare LRTI incidence in each intervention arm (Tx1 and Tx2) to LRTI in the placebo arm (Tx3). Investigators hypothesize that children less than five years old in intervention homes will experience lower LRTI.

Aim 2: Compare indoor PM2.5 concentrations in each treatment arm relative to the placebo arm. Investigators hypothesize that the intervention homes will have lower indoor PM2.5 concentrations.

Aim 3: Compare effectiveness and sustainability of treatment strategies relative to placebo, both within and between regional sites. Investigators hypothesize that Tx1 will be more effective and sustainable than Tx2.

Impact. LRTI is an important cause of morbidity among children, and exposure to biomass smoke puts children at a greater risk of LRTI. By reducing in-home wood smoke exposures, this study will evaluate sustainable evidence-based and culturally appropriate strategies for decreasing occurrence of LRTI. In addition, comparing the effectiveness of these interventions across three unique rural and Native regions will inform translation of study findings into diverse settings that utilize biomass fuels for heating and cooking.

ELIGIBILITY:
Inclusion Criteria:

* Eligible homes will be any home in the described communities that uses a wood stove as a primary heating source, and has one or more children under the age of five years. The home must include a parent who is capable and willing to record symptom data for the enrolled children and wood stove usage data.

Exclusion Criteria:

* None.

Max Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 523 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2020-03 (Actual); Study Completion 2020-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Curtis W Noonan, Ph.D., Principal Investigator — University of Montana; Tony J Ward, Ph.D., Principal Investigator — University of Montana
Locations (1):
- University of Montana, Missoula, Montana, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The KidsAIR study took place in rural areas of Alaska (AK), Navajo Nation (NN), and western Montana (WMT) where wood stoves are a common source of heating during the colder winter months. Contact with potentially eligible households occurred through clinics and advertisements. Households were enrolled from 2014 through 2018.
Units Other Than Participants: Household
Period: Overall Study
Arm/Group | Education Intervention (Tx1) | Air Filtration Unit Treatment (Tx2) | Placebo Intervention (Tx3)
Started | 176; 118 Household | 176; 115 Household | 171; 114 Household
Completed | 126; 81 Household | 123; 79 Household | 118; 78 Household
Not Completed | 50; 37 Household | 53; 36 Household | 53; 36 Household

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Education Intervention (Tx1) | Air Filtration Unit Treatment (Tx2) | Placebo Intervention (Tx3) | Total
Number analyzed (Participants) | 176 | 176 | 171 | 523
Age, Customized [Count of Participants; unit: Participants]
  < 1 year | 38 | 40 | 38 | 116
  1 - 4 years | 115 | 116 | 113 | 344
  Unknown | 24 | 20 | 20 | 64
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 70 | 65 | 64 | 199
  Male | 76 | 81 | 80 | 237
  Unknown | 30 | 30 | 27 | 87
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 7 | 2 | 14
  Not Hispanic or Latino | 146 | 146 | 149 | 441
  Unknown or Not Reported | 25 | 23 | 20 | 68
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 68 | 63 | 61 | 192
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 72 | 79 | 81 | 232
  More than one race | 11 | 12 | 9 | 32
  Unknown or Not Reported | 25 | 22 | 20 | 67
Region of Enrollment [Number; unit: participants]
  United States | 176 | 176 | 171 | 523
Received influenza vaccine [Count of Participants; unit: Participants]
  Yes | 64 | 61 | 68 | 193
  No | 81 | 83 | 76 | 240
  Unknown | 31 | 32 | 27 | 90

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With at Least One LRTI During Follow-up Period
Description: The occurrence and duration of LRTI among children will be assessed using active surveillance within the home. Identification of LRTI episodes will occur through a three step process: (1) parent reporting of symptoms; (2) Community Coordinator collection of confirmatory and severity data; and (3) physician classification of case status based on data collected by the Community Coordinator, and when available, data collected from a clinic or hospital.
Time Frame: The participants will be followed for four months during each of two successive winter periods for a total of eight months of observation.
Population: Children were evaluated during two consecutive winters for occurrence of lower respiratory tract infection (LRTI). Below are number of children with at least one LRTI during follow-up period.
Measure: Count of Participants; unit: Participants
Arm/Group | Education Intervention (Tx1) | Air Filtration Unit Treatment (Tx2) | Placebo Intervention (Tx3)
Number analyzed (Participants) | 154 | 156 | 151
Participants
  Recorded LRTI | 16 | 20 | 17
  No recorded LRTI | 138 | 136 | 134
Statistical Analysis 1: Comparison: Air Filtration Unit Treatment (Tx2) vs Placebo Intervention (Tx3); Mixed effects logistic regression model with presence of LRTI as outcome (yes or no); assigned treatment as primary exposure variable relative to placebo; adjusted for child age and person-time at-risk; nested random term: home:cohort:area. Results presented as odds ratios with 95% Confidence Intervals; Test type: Superiority; p = 0.68, Mixed Models Analysis; Odds Ratio (OR) = 1.23, 95% CI 2-sided [0.46 to 3.32] — Odds ratio for air filter treatment relative to placebo
Statistical Analysis 2: Comparison: Education Intervention (Tx1) vs Placebo Intervention (Tx3); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.96, Mixed Models Analysis; Odds Ratio (OR) = 0.98, 95% CI 2-sided [0.35 to 2.72] — Odds ratio for filter treatment relative to placebo

2. Secondary Outcome: Fine Particulate Matter Concentrations
Description: Fine particulate matter (PM2.5) concentrations by study arm
Time Frame: Six consecutive days during a four month winter period
Population: Assessment made at the household level
Measure: Mean (Standard Deviation); unit: Microgram/cubic meter
Units Other Than Participants: Household
Arm/Group | Education Intervention (Tx1) | Air Filtration Unit Treatment (Tx2) | Placebo Intervention (Tx3)
Number analyzed (Participants) | 154 | 156 | 151
Number analyzed (Household) | 84 | 84 | 85
Microgram/cubic meter | 36 (45) | 30 (37) | 32 (36)
Statistical Analysis 1: Comparison: Air Filtration Unit Treatment (Tx2) vs Placebo Intervention (Tx3); Linear mixed model with natural-log transformed 6-day mean indoor PM2.5 as outcome; assigned treatment as primary exposure variable; adjusted for child age; nested random term: cohort:area. Results presented as effect estimates with 95% Confidence Intervals and reported as percent differences in geometric mean PM2.5; Test type: Superiority; p = 0.250, Mixed Models Analysis; percent differences in geometric mean PM = -6.96, 95% CI 2-sided [-30.50 to 24.55]
Statistical Analysis 2: Comparison: Education Intervention (Tx1) vs Placebo Intervention (Tx3); [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.295, Mixed Models Analysis — Statistical significance selected as 95% confidence interval of the estimation parameter that excludes the null value, 0; percent differences in geometric mean PM = 11.77, 95% CI 2-sided [-16.57 to 49.72] — Difference in indoor PM2.5 for education treatment versus placebo

ADVERSE EVENTS:
Time Frame: The participants will be followed for four months during each of two successive winter periods for a total of eight months of observation.
Arm/Group | Education Intervention (Tx1) | Air Filtration Unit Treatment (Tx2) | Placebo Intervention (Tx3)
All-Cause Mortality (participants affected / at risk) | 0/176 | 0/176 | 0/171
Serious Adverse Events (participants affected / at risk) | 0/176 | 0/176 | 0/171
Other Adverse Events (participants affected / at risk) | 0/176 | 0/176 | 0/171

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-11-11): https://cdn.clinicaltrials.gov/large-docs/34/NCT02240134/Prot_SAP_000.pdf